CLINICAL TRIAL: NCT02586298
Title: Autologous Mitochondrial Transfer as a Complementary Technique to ICSI to Improve Oocyte and Embryo Quality in IVF Patients. Pilot Study
Brief Title: Autologous Mitochondrial Transfer in ICSI to Improve Oocyte and Embryo Quality in IVF Patients. Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1501-VLC-005-AP
Record Dates: First submitted 2015-10-21; First posted 2015-10-26 (Estimated); Last update posted 2017-08-23 (Actual); Status verified 2017-08

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Sperm Injections, Intracytoplasmic

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- ICSI with mitochondria (Experimental): Half of the Metaphase II oocytes retrieved after the controlled ovarian stimulation will be randomized to this group and autologous mitochondria from the patient's ovarian cortex will be introduced into the oocyte during the intracytoplasmic sperm injection in the vitro fertilization treatment.
  Interventions: Other: Autologous mitochondria with ICSI
- Control ICSI without mitochondria (Active Comparator): The other half of the metaphase II oocytes retrieved after the controlled ovarian stimulation will be randomized to this group and will not receive autologous mitochondria during the intracytoplasmic sperm injection (ICSI) in the vitro fertilization treatment. Control Group
  Interventions: Other: STANDARD ICSI PROCEDURE

INTERVENTIONS:
Other: Autologous mitochondria with ICSI — Autologous mitochondria during the intracytoplasmic sperm injection (ICSI) process will be added to this randomized group of oocytes.
  Arms: ICSI with mitochondria
Other: STANDARD ICSI PROCEDURE — STANDARD ICSI PROCEDURE
  Arms: Control ICSI without mitochondria

SUMMARY:
The principle objective is to improve embryo quality through autologous micro-injection of mitochondria isolated from Ovarian stem cells into the oocytes themselves, as a complementary ICSI technique in patients with low embryo quality in previous IVF cycles and in those who did not bear children.

This improvement in embryo quality will be determined through on-going pregnancy rate after treatment and/or improvement in embryo quality according to morphological (ASEBIR-"Association for the study of Biology in Reproductive Science), morphokinetic criteria and in Preimplantation Genetic Screening.

Using an adaptive design, retrieved oocytes of approximately 60 patients will be randomized in the first part of the study to two treatment groups; standard ICSI procedure without mitochondrial supplementation and ICSI with autologous mitochondrial supplementation. Following an interim analysis of outcomes, an additional 130 patients may be added, for a total of 190 patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients must have read, understood and signed the ICF.
* Age ≤ 42 years.
* Serum AMH ≥ 4 pM/L.
* Previous IVF cycle with 5 or more metaphase II oocytes after retrieval
* BMI < 30.
* Will undergo an IVF cycle with arrays in Preimplantation Genetic Screening.
* Semen sample with concentrations exceeding 3 million/mL progressive motile sperm.

Present with a history of at least one previous cycle of IVF with embryo transfer and no pregnancy due to low embryo quality. Low embryo quality is understood as > 70% of the embryos obtained being included in the worst prognosis category according to any of the following criteria:

1. Low or abnormal Fertilization Rate despite semen count > 3 million/mL.
2. Deficient quality embryos according to morphological criteria established by ASEBIR:

   i. Embryo D2 and D3: classified as Type C or Type D according to ASEBIR criteria.

   ii. Embryo D5 or blastocyst: Inner cell mass absent, with few cells and difficult differentiation, Trophectoderm with very few cells. Type C or D of ASEBIR.
3. Embryos of deficient quality according to morphokinetic criteria established (28) for EmbryoScope Time-Lapse if this incubator has been used.

   i.Category 4: Embryos of 1 or 2 pronuclei (PN) formed from 1 to 2 cells at 27h, from 2 to 6 cells on D2 and 4 or >8 cells or morula on D3. The embryo can present with asymmetrical and multinucleated blastomeres. Degree of fragmentation < 50%.

   ii. Category 5: Embryo with any number of cells at 27h, on D2 and D3. Asymmetrical, multinucleated blastomeres and any degree of fragmentation. Atretic embryos and those with arrested embryo development belong to this category.
4. All cases without embryo transfer due to any chromosomal abnormality detected through PGD or PGS techniques.
5. All cases without transfer due to the presence of embryos that present a blockage of embryo development before D3.

If the morphological quality criteria established under points 2, 3 and 4 give contradictory results, the result obtained through PGD/PGS (point 4) will prevail over the morphokinetic parameters (point 3) and this, in turn, will prevail over the classic morphological criteria (point 2).

Exclusion Criteria:

* Formal contraindication for ovarian cortex biopsy or follicle puncture.
* Severe male factor (concentration<3 million/mL of progressive motile sperm).
* Any characteristic incompatible with carrying out a new IVF cycle at IVI Valencia.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Rate of ongoing pregnancy | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Elena Labarta, MD PhD, Study Director — Gynecologist Specialist TRA, IVI Valencia; Antonio Pellicer, MD PhD, Principal Investigator — Gynecologist specialist TRA, President IVI Valencia
Locations (1):
- IVI Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Labarta E, de Los Santos MJ, Herraiz S, Escriba MJ, Marzal A, Buigues A, Pellicer A. Autologous mitochondrial transfer as a complementary technique to intracytoplasmic sperm injection to improve embryo quality in patients undergoing in vitro fertilization-a randomized pilot study. Fertil Steril. 2019 Jan;111(1):86-96. doi: 10.1016/j.fertnstert.2018.09.023. Epub 2018 Nov 24. PMID 30477915